CLINICAL TRIAL: NCT04483973
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety and Efficacy of SPI-1005 in Severe COVID-19 Patients
Brief Title: SPI-1005 Treatment in Severe COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1005-292
Record Dates: First submitted 2020-07-13; First posted 2020-07-23 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Coronavirus; Coronavirus Infection; Corona Virus Infection
Keywords: ebselen; SPI-1005; COVID-19; Covid; SARS-COV-2; Mpro; main protease; PLpro; papain-like protease
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SPI-1005 400 mg BID (Experimental): Oral administration of SPI-1005 400 mg BID for 14 days, with 30-day follow-up
  Interventions: Drug: Ebselen
- SPI-1005 800 mg BID (Experimental): Oral administration of SPI-1005 800 mg BID for 14 days, with 30-day follow-up
  Interventions: Drug: Ebselen
- Placebo (Placebo Comparator): Oral administration of matching placebo BID for 14 days, with 30-day follow-up
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ebselen — Glutathione peroxidase mimetic
  Other Names: SPI-1005
  Arms: SPI-1005 400 mg BID; SPI-1005 800 mg BID
Drug: Placebo — Matching placebo containing excipients
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, dose escalation, multi-center clinical trial (RCT) of SPI-1005 in adult subjects with positive PCR test for novel SARS-CoV-2 (nCoV2) and severe symptoms of COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Positive nCoV2 PCR test by nasopharyngeal, oral, saliva, or respiratory sample
* Clinical signs, symptoms, and respiratory status consistent with severe COVID-19
* Score of 5-7 on the WHO Ordinal Scale
* Onset of severe COVID-19 symptoms ≤7 days of study enrollment
* Subject is in-patient at time of randomization to study treatment
* Subject or legally authorized representative is willing and able to provide informed consent, and agrees for subject to comply with planned study procedures including reproductive requirements

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding.
* Participation in another interventional investigational drug or device study concurrently or within 30 days prior to study consent.
* Patients with impaired hepatic or renal function.
* Subject has any other illness or condition that, in the opinion of the investigator, would prohibit the subject from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 30 days

SECONDARY OUTCOMES:
WHO Ordinal Scale | 30 days
  Clinical outcome assessed by WHO Ordinal Scale for Clinical Improvement. Scale is 0-8 where higher score is worse outcome.
Degree of supplemental oxygen | 30 days
  Respiratory status assessed by degree of supplemental oxygen (e.g. mask oxygen, mechanical ventilation)
Peripheral Oxygen Saturation (SpO2) | 30 days
  Peripheral oxygen saturation measured by pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, Principal Investigator — Yale University
Locations (7):
- United States (7):
  - Yale University, New Haven, Connecticut
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Kansas University Medical Center, Kansas City, Kansas
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jin Z, Du X, Xu Y, Deng Y, Liu M, Zhao Y, Zhang B, Li X, Zhang L, Peng C, Duan Y, Yu J, Wang L, Yang K, Liu F, Jiang R, Yang X, You T, Liu X, Yang X, Bai F, Liu H, Liu X, Guddat LW, Xu W, Xiao G, Qin C, Shi Z, Jiang H, Rao Z, Yang H. Structure of Mpro from SARS-CoV-2 and discovery of its inhibitors. Nature. 2020 Jun;582(7811):289-293. doi: 10.1038/s41586-020-2223-y. Epub 2020 Apr 9. PMID 32272481
- [Background] Menendez CA, Bylehn F, Perez-Lemus GR, Alvarado W, de Pablo JJ. Molecular characterization of ebselen binding activity to SARS-CoV-2 main protease. Sci Adv. 2020 Sep 11;6(37):eabd0345. doi: 10.1126/sciadv.abd0345. Print 2020 Sep. PMID 32917717
- [Background] Weglarz-Tomczak E, Tomczak JM, Talma M, Burda-Grabowska M, Giurg M, Brul S. Identification of ebselen and its analogues as potent covalent inhibitors of papain-like protease from SARS-CoV-2. Sci Rep. 2021 Feb 11;11(1):3640. doi: 10.1038/s41598-021-83229-6. PMID 33574416
- [Background] Brown AS, Ackerley DF, Calcott MJ. High-Throughput Screening for Inhibitors of the SARS-CoV-2 Protease Using a FRET-Biosensor. Molecules. 2020 Oct 13;25(20):4666. doi: 10.3390/molecules25204666. PMID 33066278
- [Background] Haritha CV, Sharun K, Jose B. Ebselen, a new candidate therapeutic against SARS-CoV-2. Int J Surg. 2020 Dec;84:53-56. doi: 10.1016/j.ijsu.2020.10.018. Epub 2020 Oct 23. No abstract available. PMID 33120196
- [Background] Chen T, Fei CY, Chen YP, Sargsyan K, Chang CP, Yuan HS, Lim C. Synergistic Inhibition of SARS-CoV-2 Replication Using Disulfiram/Ebselen and Remdesivir. ACS Pharmacol Transl Sci. 2021 Mar 26;4(2):898-907. doi: 10.1021/acsptsci.1c00022. eCollection 2021 Apr 9. PMID 33855277
- [Background] Sies H, Parnham MJ. Potential therapeutic use of ebselen for COVID-19 and other respiratory viral infections. Free Radic Biol Med. 2020 Aug 20;156:107-112. doi: 10.1016/j.freeradbiomed.2020.06.032. Epub 2020 Jun 26. PMID 32598985